CLINICAL TRIAL: NCT04949997
Title: Evaluation of Left Ventricular Systolic Function in Heart Failure With Middle Ejection Fraction by 3D Speckle Tracking Imaging
Brief Title: Evaluation of Systolic Function in Heart Failure With Middle Ejection Fraction by 3D Speckle Tracking Imaging
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2017152
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
Keywords: median ejection fraction; 3D-STI
MeSH Terms: conditions — Heart Failure | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: patients without heart failure
- HF: patients with heart failure
  Interventions: Other: diagnose

INTERVENTIONS:
Other: diagnose — HF was divided into HF with preserved ejection fraction, HF with median ejection fraction and HF with reduced ejection fraction.
  Groups: HF

SUMMARY:
In 2016, the European Heart Association defined the median ejection fraction heart failure for the first time. More research is needed to improve our understanding of this population, so as to make the best clinical decision and improve the prognosis. In this study, 3D-STI was used to evaluate left ventricular systolic function in heart failure with median ejection fraction.

DETAILED DESCRIPTION:
As the final manifestation of cardiovascular disease and the main cause of death, heart failure is one of the important challenges threatening human health in the 21st century. In 2016, the European Heart Association proposed a new classification standard for heart failure. In particular, for the first time, heart failure with median ejection fraction has been clearly defined. These patients have received more and more attention, but there are still relatively few studies on them. More research is needed to improve our understanding of this part of the population in order to make the best clinical decisions and improve the prognosis. 3D speckle tracking technology is a new technology developed on the basis of real-time three-dimensional echocardiography and speckle tracking technology. It is gradually recognized in the evaluation of left ventricular systolic and diastolic function, especially in the evaluation of cardiotoxicity of chemotherapy drugs. At present, the application of 3D-STI in the evaluation of left ventricular systolic function in heart failure with median ejection fraction is limited and needs further study.In this study, 3D-STI was used to evaluate left ventricular systolic function in heart failure with median ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

Meeting the diagnostic and classification criteria of heart failure proposed in the 2016 ESC guidelines for the diagnosis and treatment of acute / chronic heart failure

Exclusion Criteria:

1. acute or chronic infectious diseases;
2. COPD, chronic bronchitis, emphysema and other serious lung diseases;
3. Autoimmune diseases;
4. Malignant tumor;
5. Acute, chronic liver disease or other reasons lead to abnormal liver function (transaminase is more than 3 times of normal value);
6. Acute and chronic kidney disease, end-stage renal disease (serum creatinine > 220 μmol/L, or creatinine clearance rate < 30 ml/min);
7. Heart valve disease;
8. Severe arrhythmia;
9. The image quality of echocardiography was poor when it was larger than three sections;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients meet the diagnostic and classification criteria of heart failure proposed in the 2016 ESC guidelines for HF but not the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
3D-STI measurement indexes | one week
  strain values of different sections from 3D-STI

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No